CLINICAL TRIAL: NCT01963182
Title: Phase II Study: Individualization of Dosage of Irinotecan in the FOLFIRI According to the Genetic Polymorphism of UGT1A1 in the First Line Treatment of Metastatic Colorectal Cancer
Brief Title: Individualization of Dosage of Irinotecan in the FOLFIRI According to the Genetic Polymorphism of UGT1A1 in the First Line Treatment of Metastatic Colorectal Cancer
Acronym: IriGen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-001275-21
Record Dates: First submitted 2013-10-10; First posted 2013-10-16 (Estimated); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: First Line Metastatic Colorectal Cancer
MeSH Terms: interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- irinotecan dose based on genetic polymorphism of UGT1A1 (Experimental)
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Irinotecan

SUMMARY:
This prospective, non randomized multicenter phase II study, will determine the feasibility of individualized dose of irinotecan with the UGT1A1 polymorphism, in patients with metastatic colorectal cancer treated with FOLFIRI.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer histologically or cytologically proven
* Indication of treatment according to the FOLFIRI + / - bevacizumab or cetuximab or panitumumab
* Age> 18 years
* Presence of at least one measurable target by RECIST
* Life expectancy> 3 months
* Satisfactory biological functions (renal, hepatic and hematologic)
* Affiliation to a social security scheme (or be the beneficiary of such a plan) under the terms of the Act of August 9, 2004
* Patient has signed, after informing the informed consent form

Exclusion Criteria:

* Patients of childbearing age and not using effective contraception during treatment and for at least three months after the end of treatment with irinotecan and at least six months after the end of treatment with bevacizumab, cetuximab or panitumumab and patient pregnant or nursing
* Patient with another pathology deemed incompatible with the entry in the protocol
* Prior treatment in metastatic
* Patients taking antiepileptic
* Allergic reaction or intolerance to irinotecan
* Heart failure , kidney , bone marrow , liver or respiratory
* Higher bilirubin 1.5 times the upper limit of normal
* Significant psychiatric or neurological abnormality
* Infectious syndrome requiring treatment with antibiotics or antiviral long-term
* Patients with chronic inflammatory bowel disease and / or bowel obstruction
* Contraindication Association St. John's wort and yellow fever vaccine
* Against Heart indication 5-FU
* Concurrent treatment with a drug test , participation in a clinical trial within <30 days
* Patient refused to sign the consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-10; Primary Completion 2019-12 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
severe toxicity (according to NCI-CTC cotation) and response with adapted dose of irinotecan | during the treatment (an expected average of 7 months)

SECONDARY OUTCOMES:
Study of the blood concentration (pharmacokinetic) of irinotecan, the SN38 and SN38-G, and bevacizumab | during the first 24 hours of the first cure
evaluation of treatment efficacy (progression-free survival, duration of response) | to progression (1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Hervé DEVAUD, MD, Principal Investigator — Centre Jean Perrin
Locations (3):
- France (3):
  - Clinique de la Châtaigneraie, Beaumont
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU Estaing, Clermont-Ferrand

REFERENCES:
- [Derived] Ginzac A, Thivat E, Petorin C, Richard D, Herviou P, Molnar I, Devaud H, Creveaux I, Ferrer F, Authier N, Jary M, Pezet D, Durando X. A phase-II study based on dose adjustment according to UGT1A1 polymorphism: is irinotecan underdosed in first-line FOLFIRI regimen for mCRC? Cancer Chemother Pharmacol. 2024 Mar;93(3):225-236. doi: 10.1007/s00280-023-04603-x. Epub 2023 Nov 7. PMID 37932443